CLINICAL TRIAL: NCT06070259
Title: Examining Patient Involvement Patterns and Trends in Participation in Bone Cancer Clinical Trials
Brief Title: Insights Into Participating in Studies for Bone Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 72278769
Record Dates: First submitted 2023-09-30; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Bone Cancer
Keywords: Bone Cancer
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical studies, with a distinct focus on bone cancer, play a crucial role in evaluating the safety and effectiveness of novel treatments for this disease. These trials serve as instrumental means to determine whether new medications surpass conventional therapies, providing substantial evidence for their broader adoption.

The primary objective is to meticulously scrutinize trial completion rates and voluntary withdrawals within this specific patient group.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Diagnosis of bone cancer
* No prior treatment for bone cancer

Exclusion Criteria:

* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Enrolled in another research study
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bone cancer patients who are actively considering enrolling in a clinical trial for the said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a bone cancer clinical research. | 3 months
Number of bone cancer study participants who remain in clinical study until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ventura C, Nunez SV, Goncalves A, Abreu C, Costa L. Bone Health in Metastatic Cancer. Semin Oncol Nurs. 2022 Apr;38(2):151278. doi: 10.1016/j.soncn.2022.151278. Epub 2022 Apr 15. PMID 35431084
- [Background] Porta-Sales J, Garzon-Rodriguez C, Llorens-Torrome S, Brunelli C, Pigni A, Caraceni A. Evidence on the analgesic role of bisphosphonates and denosumab in the treatment of pain due to bone metastases: A systematic review within the European Association for Palliative Care guidelines project. Palliat Med. 2017 Jan;31(1):5-25. doi: 10.1177/0269216316639793. Epub 2016 Jul 10. PMID 27006430
- [Background] Niiyama Y, Kawamata T, Yamamoto J, Furuse S, Namiki A. SB366791, a TRPV1 antagonist, potentiates analgesic effects of systemic morphine in a murine model of bone cancer pain. Br J Anaesth. 2009 Feb;102(2):251-8. doi: 10.1093/bja/aen347. Epub 2008 Nov 26. PMID 19038965

DOCUMENTS (1):
  • Informed Consent Form (2023-09-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT06070259/ICF_000.pdf